CLINICAL TRIAL: NCT04949152
Title: Brazilian Diabetes Study: a Type 2 Diabetes Prospective Cohort
Acronym: BDS
Status: Recruiting | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, MD, PhD, University of Campinas, Brazil
Other Study IDs: 41618915.1.0000.5404
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Diseases; Diabete Mellitus; Coronary Artery Disease
Keywords: diabetes; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ongoing prospective cohort of type 2 diabetes individuals.

DETAILED DESCRIPTION:
The study population included individuals with type 2 diabetes aged between 40 and 70 years old, living in the metropolitan area of Campinas, Brazil. The volunteers were recruited between 2016 and 2020 through radio, newspaper, television and social media advertisements. A total of 1046 participants were enrolled into the study so far.

All participants were firstly invited to an interview with the physician-researcher for medical story register and physical examination. Afterwards, all participants were submitted to the following procedures: blood and urine samples collection, dual-energy X-ray absorptiometry, 6 minutes walk test, hand strength test, bone densitometry test, diabetic polyneuropathy evaluation, advanced glycation end-product measurement, electrocardiogram, echocardiogram, carotid doppler ultrasound, flow-mediated dilation, diabetic retinopathy assessment, ambulatory blood pressure monitoring and cardiac computed tomography for calcium scoring. After full examination, patients were contacted every year for 5 years for endpoints registration. The primary endpoint was a composite of all-cause mortality, myocardial infarction, stroke and myocardial revascularization. Secondary endpoints were end-stage kidney disease requiring dialysis and limb amputation. Study data were collected and managed using REDCap electronic data capture tools.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 diabetes
* Age between 40 and 70 years old

Exclusion Criteria:

* Unconfirmed diagnosis of diabetes
* Intellectual disability

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals from both genders, aged 40 to 70 years-old, with confirmed diagnosis of type 2 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 1046 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 5 years
  All cause death, myocardial infarction, stroke, myocardial revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical research center, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barreto J, Chaves F, Fernandes VHR, Jesus DC, Nascimento MA, Lira RPC, Nadruz W, Arieta C, Sposito AC. Proteinuria in early referral to spectral domain optical coherence tomography for macular edema detection in type 2 diabetes individuals: results from the Brazilian diabetes study. Curr Med Res Opin. 2022 Dec;38(12):2141-2148. doi: 10.1080/03007995.2022.2131302. Epub 2022 Nov 4. PMID 36190762
- [Derived] Barreto J, Wolf V, Bonilha I, Luchiari B, Lima M, Oliveira A, Vitte S, Machado G, Cunha J, Borges C, Munhoz D, Fernandes V, Kimura-Medorima ST, Breder I, Fernandez MD, Quinaglia T, Oliveira RB, Chaves F, Arieta C, Guerra-Junior G, Avila S, Nadruz W, Carvalho LSF, Sposito AC; Brazilian Heart Study Group. Rationale and design of the Brazilian diabetes study: a prospective cohort of type 2 diabetes. Curr Med Res Opin. 2022 Apr;38(4):523-529. doi: 10.1080/03007995.2022.2043658. Epub 2022 Mar 2. PMID 35174749